CLINICAL TRIAL: NCT01185717
Title: Epidemiology of Anti-JCV Antibody Prevalence in Multiple Sclerosis Patients
Brief Title: JC-virus (JCV) Epidemiology in Multiple Sclerosis (MS)
Acronym: JEMS
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 100JC401
Record Dates: First submitted 2010-08-19; First posted 2010-08-20 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the study is to estimate the prevalence of anti-JCV antibodies in multiple sclerosis (MS) participants.

DETAILED DESCRIPTION:
This is a cross-sectional, multi-center, multi-national, epidemiological study to estimate the prevalence of anti-JCV antibody in MS participants. This study will provide an estimate of the prevalence of anti-JCV antibody in the MS population and will investigate inter-country differences.

ELIGIBILITY:
Key Inclusion Criteria:

* All candidates for this study must have the ability to understand the purpose of the study and provide signed and dated informed consent.
* All patients with a diagnosis of Multiple Sclerosis (MS) of any type, irrespective of their treatment, are eligible to participate once.

Key Exclusion Criteria:

* None

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Multiple Sclerosis (MS) patients will be enrolled in Europe, Canada, and Australia.
  Patient enrollment from each country will be commensurate with the distribution of MS patients among all participating countries.
Sampling Method: Non-Probability Sample
Enrollment: 7726 (Actual)
Dates: Start 2010-09; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of anti-JCV antibodies | Single timepoint (Day 1)
  Prevalence of anti-JCV antibodies will be estimated as the number of participants with anti-JCV antibodies detected in serum divided by the total number of participants with a serum sample that was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen

REFERENCES:
- [Background] da Silva AM, Santos ME; Portuguese JEMS Study Investigators. JCV epidemiology in MS (JEMS)--epidemiology of anti-JCV antibody prevalence in multiple sclerosis patients--Portuguese data. J Neurol Sci. 2014 Feb 15;337(1-2):119-22. doi: 10.1016/j.jns.2013.11.031. Epub 2013 Dec 1. PMID 24369270